CLINICAL TRIAL: NCT02178267
Title: Effect Of Probiotics On Resistant Bacteria Colonization Preterm Newborn Infants Receiving Antibiotics In Neonatal Intensive Care Unit
Brief Title: Probiotics On Resistant Bacteria Colonization In Preterm Receiving Antibiotics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baskent University (Other)
Responsible Party: Principal Investigator, Dr Abdullah Kurt, Neonatologist, Baskent University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: Kurt - 1
Record Dates: First submitted 2014-06-13; First posted 2014-06-30 (Estimated); Last update posted 2014-06-30 (Estimated); Status verified 2014-06

CONDITIONS: Infant, Premature, Diseases
Keywords: Newborn, preterm, probiotic, resistant microorganisms
MeSH Terms: conditions — Infant, Premature, Diseases; Premature Birth

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Lactobacillus reuteri (Experimental): The study was performed by two groups. And these groups were constituted from the newborn preterm infants who are received probiotics (Lactobacillus reuteri) and no probiotics.
  Interventions: Dietary Supplement: Lactobacillus reuteri (biogai AB, Sweden)

INTERVENTIONS:
Dietary Supplement: Lactobacillus reuteri (biogai AB, Sweden) — Lactobacillus reuteri (biogai AB, Sweden) was given to probiotic group, same way to all newborn newborn preterm infants, directly oral feeding and without any along with a mixture, admission following the in nicu, as a daily dose 1x108 cfu / day (1x5 drops / day) during hospitalization
  Other Names: Probiotics were randomly given to newborn preterm infants.

SUMMARY:
In this study, the investigators investigated the effect of probiotic use on colonization of resistant microorganisms in newborn preterm infants receiving antibiotics. This study of the use of probiotics in preterm neonates in neonatal intensive care units expect to prevent colonization by resistant microorganisms.

DETAILED DESCRIPTION:
The gut which is sterile in newborn preterm infants begins to colonize with birth. Factors such as developmental immaturity of the immune system, encountering with the flora of neonatal intensive care unit, exposure to diagnostic and therapeutic interventional procedures, use of antibiotics, delay of enteral feeding may poorly affect the development of natural and mucosal immunity of intestine in newborns preterm during postnatal period. Exposure to these factors, newborn preterm infants' life threatens especially to change the development of the normal intestinal flora and intestinal immunity. Many randomized controlled studies reported that probiotics reduce intestinal inflammatory process and prevent colonization with pathogenic microorganisms of the intestines . In this study, the investigators investigated the effect of probiotic use on colonization of resistant microorganisms in newborn preterm infants receiving antibiotics.

ELIGIBILITY:
Inclusion Criteria:

* The study were included ≤36 weeks gestational age newborn preterm infants requiring antibiotic treatment and/or prophylaxis.

Exclusion Criteria:

* Newborn preterm infants who are congenital anomalies and not require antibiotic therapy and undergoing intestinal operation were excluded from the study.

Ages: 1 Day to 28 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 51 (Actual)
Dates: Start 2011-01; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
The use of probiotics in newborn preterm infants receiving antibiotics will be investigated type of resistant microorganisms in the flora of intestinal and nasal. | Up to 12 month
  The gut which is sterile in newborn preterm infants begins to colonize with birth. Factors such as developmental immaturity of the immune system, encountering with the flora of neonatal intensive care unit, exposure to diagnostic and therapeutic interventional procedures, use of antibiotics, delay of enteral feeding may poorly affect the development of natural and mucosal immunity of intestine in newborns preterm during postnatal period. Exposure to these factors, newborn preterm infants' life threatens especially to change the development of the normal intestinal flora and intestinal immunity. Many randomized controlled studies reported that probiotics reduce intestinal inflammatory process and to prevent colonization with pathogenic microorganisms of the intestines . In this study, we investigated the effect use of probiotic on colonization of resistant microorganisms in newborn preterm infants receiving antibiotics.

SECONDARY OUTCOMES:
Types Of Resistant Microorganisms In The Culture | Up to 12 month
  In the culture, all possible resistant microorganisms such as methicillin-resistant Staphylococci aureus, Enterococcus, Klebsiella spp, Escherichia coli, Pseudomonas aeruginosa, Enterobacter, Acinetobacter, Serratia, Candida species were investigated.

CONTACTS AND LOCATIONS:
Overall Officials: Abdullah Kurt, Neonatology, Principal Investigator — Baskent University